CLINICAL TRIAL: NCT05875909
Title: Corneal Flap Transplantation for Macular Hole Repair of High Myopia
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-025
Record Dates: First submitted 2023-05-17; First posted 2023-05-25 (Actual); Last update posted 2023-05-25 (Actual); Status verified 2023-04

CONDITIONS: Retinal Perforations; Myopia, Degenerative
Keywords: corneal flap transplantation; femtosecond laser small incision lenticule extraction; macular hole; surgical technique
MeSH Terms: conditions — Retinal Perforations; Myopia, Degenerative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- corneal flap transplantation (Experimental): Patients with macular holes underwent a 25-gauge, 3-port pars plana vitrectomy . Fluid-air exchange was performed in patients with pathologic myopia suffering from macular holes with retinal detachment. We used a flute needle to drain the subretinal fluid. A corneal flap was obtained by small incision lenticule extraction (SMILE). Stripping pliers were applied to spread corneal flap over the macular hole. A drop of fresh autologous whole blood was dripped over the corneal flap to immobilise it. The vitreous cavity was filled with 14% perfluoropropane (C3F8) for macular holes with retinal detachment . The surgical incision was self-closed or sutured with a 6-0 polyglactin 910 suture . The patients were instructed to maintain a prone position for 2 weeks postoperatively.
  Interventions: Procedure: corneal flap transplantation

INTERVENTIONS:
Procedure: corneal flap transplantation — Patients with macular holes underwent a 25-gauge, 3-port pars plana vitrectomy . Fluid-air exchange was performed in patients with pathologic myopia suffering from macular holes with retinal detachment. We used a flute needle to drain the subretinal fluid. A corneal flap was obtained by small incision lenticule extraction (SMILE). Stripping pliers were applied to spread corneal flap over the macular hole. A drop of fresh autologous whole blood was dripped over the corneal flap to immobilise it. The vitreous cavity was filled with 14% perfluoropropane (C3F8) for macular holes with retinal detachment . The surgical incision was self-closed or sutured with a 6-0 polyglactin 910 suture . The patients were instructed to maintain a prone position for 2 weeks postoperatively.

SUMMARY:
The goal of this clinical trial is to learn about an innovative surgical technique for macular hole repair. This technique is for patients with high myopia using pars plana vitrectomy (PPV) combined with corneal flap transplantation. The main questions it aims to answer are:

* Is the innovative surgical technique useful for patients?
* Is the surgical technique safe for patients?

Participants will:

* Undergo PPV combined with corneal flap transplantation to cover the macular hole.
* Maintain a prone position for 2 weeks postoperatively.
* Be observed by visual acuity, slit lamp, optical coherence tomography (OCT) and fundus photography for 1 year after surgery.

DETAILED DESCRIPTION:
We describe an innovative surgical technique for macular hole repair using pars plana vitrectomy (PPV) combined with corneal flap transplantation. The corneal flap was sealed with autologous blood. The vitreous cavity was then filled with perfluoropropane (C3F8) or sterile air.

ELIGIBILITY:
Inclusion Criteria:

* Patients with macular hole and retinal detachment caused by pathologic myopia.

Exclusion Criteria:

* Patients with previous retinal surgery, trauma, other ocular diseases that could affect the vision, for example choroidal neovascularization, diabetic retinopathy, or opaque corneas were excluded.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-02-23 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
best-corrected visual acuity | one month to one year after surgery
  the best-corrected visual acuity of the patients after surgery
complications | one month to one year after surgery
  inflammation, infection, rejection reaction, ocular hypertension, ocular hypotension, recrudescent macular hole, parafoveal atrophy, corrugations or irregularities, choroidal neovascularisation, retinal detachment, cystoid macular oedema, reactive pigment epithelial hyperplasia, displacement, or opacification of the corneal flap
closure of the macular holes | one month to one year after surgery
  closure of the macular holes observed using optical coherence tomography
reattachment of the retina | one month to one year after surgery
  reattachment of the retina observed using optical coherence tomography

CONTACTS AND LOCATIONS:
Overall Officials: Yongping Hu, MD, Study Chair — Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, China
Locations (1):
- Department of Ophthalmology, Affiliated Hangzhou First People's Hospital, Zhejiang University School of Medicine, Hangzhou, China, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No
The data will be used as part of other studies.

REFERENCES:
- [Background] Zhu K, Lei B, Wong W, Zhang J, Guo Y, Chen H, Song F, Chang Q, Xu G, Zhang Y. COMPARISON OF THE INTERNAL LIMITING MEMBRANE INSERTION TECHNIQUE AND THE INVERTED INTERNAL LIMITING MEMBRANE FLAP TECHNIQUE WITH VITRECTOMY TO TREAT MACULAR HOLE-ASSOCIATED RETINAL DETACHMENT. Retina. 2021 Jan 1;41(1):37-44. doi: 10.1097/IAE.0000000000002804. PMID 32310627
- [Background] Ling L, Liu Y, Zhou B, Gao F, Hu Z, Tian M, Xing Y, Ji K, Sun T, Zhou W. Inverted Internal Limiting Membrane Flap Technique versus Internal Limiting Membrane Peeling for Vitrectomy in Highly Myopic Eyes with Macular Hole-Induced Retinal Detachment: An Updated Meta-Analysis. J Ophthalmol. 2020 Aug 24;2020:2374650. doi: 10.1155/2020/2374650. eCollection 2020. PMID 32908680
- [Background] Peng J, Chen C, Zhang H, Zhang L, Liu J, Ren J, Zhao P. LONG-TERM SURGICAL OUTCOMES OF LENS CAPSULAR FLAP TRANSPLANTATION IN THE MANAGEMENT OF REFRACTORY MACULAR HOLE. Retina. 2021 Apr 1;41(4):726-734. doi: 10.1097/IAE.0000000000002922. PMID 32732611
- [Background] Yadav NK, Venkatesh R, Thomas S, Pereira A, Shetty KB. Novel Method of Plugging the Hole: Anatomical and Functional Outcomes of Human Amniotic Membrane-Assisted Macular Hole Surgery. J Curr Ophthalmol. 2020 Dec 12;32(4):361-367. doi: 10.4103/JOCO.JOCO_189_20. eCollection 2020 Oct-Dec. PMID 33553838
- [Background] Takeuchi J, Kataoka K, Shimizu H, Tomita R, Kominami T, Ushida H, Kaneko H, Ito Y, Terasaki H. INTRAOPERATIVE AND POSTOPERATIVE MONITORING OF AUTOLOGOUS NEUROSENSORY RETINAL FLAP TRANSPLANTATION FOR A REFRACTORY MACULAR HOLE ASSOCIATED WITH HIGH MYOPIA. Retina. 2021 May 1;41(5):921-930. doi: 10.1097/IAE.0000000000003000. PMID 33079787
- [Background] Chen SN, Yang CM. Perfluorocarbon Liquid-Assisted Neurosensory Retinal Free Flap for Complicated Macular Hole Coexisting with Retinal Detachment. Ophthalmologica. 2019;242(4):222-233. doi: 10.1159/000502443. Epub 2019 Sep 18. PMID 31533121
- [Background] Tsai DC, Huang YH, Chen SJ. Parafoveal atrophy after human amniotic membrane graft for macular hole in patients with high myopia. Br J Ophthalmol. 2021 Jul;105(7):1002-1010. doi: 10.1136/bjophthalmol-2019-315603. Epub 2020 Jul 31. PMID 32737034
- [Background] Li M, Tang J, Jia Z, Yao Y, Jin E, Wang Z, Hu J, Sun G, Yin H, Liang J, Li X, Jiang Y, Qu J, Zhao M. Long-term follow-up of primary silicone oil tamponade for retinal detachment secondary to macular hole in highly myopic eyes: a prognostic factor analysis. Eye (Lond). 2021 Feb;35(2):625-631. doi: 10.1038/s41433-020-0922-0. Epub 2020 May 6. PMID 32376975
- [Background] Lyu J, Xia F, Zhao P. Intraoperative Perfluorocarbon Liquid Tamponade Technique for Treatment of Extensive Retinal Detachment Secondary to a Myopic Macular Hole. Retina. 2023 Apr 1;43(4):698-704. doi: 10.1097/IAE.0000000000003429. Epub 2023 Mar 22. PMID 35174806